CLINICAL TRIAL: NCT03547115
Title: Phase 1, Open-label, Study of Voruciclib in Subjects With Relapsed and/or Refractory B Cell Malignancies or AML After Failure of Prior Standard Therapies and Voruciclib in Combination With Venetoclax in Subjects With Relapsed/Refractory AML
Brief Title: A Study of Voruciclib Alone or in Combination With Venetoclax in Subjects With B-Cell Malignancies or AML
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: MEI Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ME-522-001
Record Dates: First submitted 2018-05-24; First posted 2018-06-06 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Follicular Lymphoma (FL); Mantle Cell Lymphoma (MCL); Marginal Zone Lymphoma (MZL); Small Lymphocytic Lymphoma (SLL); Chronic Lymphocytic Leukemia (CLL); Diffuse Large B-cell Lymphoma (DLBCL); Acute Myeloid Leukemia (AML)
Keywords: B-Cell Malignancies, AML, voruciclib, venetoclax, CDK Inhibitor
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Large B-Cell, Diffuse; Leukemia, Myeloid, Acute | interventions — voruciclib; venetoclax

STUDY DESIGN:
Intervention Model Description: This is a Phase 1, open-label, 3 + 3 dose escalation study to determine the safety and preliminary efficacy of voruciclib alone or in combination with venetoclax.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- voruciclib monotherapy and voruciclib in combination with venetoclax (Experimental): voruciclib monotherapy - Open-label, 3 + 3 dose escalation study which may enroll up to 6 subjects at each dose level and disease type (AML or B-cell malignancies)
  voruciclib and venetoclax - Open-label, 3 + 3 dose escalation study which may enroll up to 6 subjects at each dose level for AML subjects
  Interventions: Drug: voruciclib monotherapy; Drug: voruciclib and venetoclax

INTERVENTIONS:
Drug: voruciclib monotherapy — Voruciclib will be administered orally
  Other Names: ME-522
Drug: voruciclib and venetoclax — Voruciclib and Venetoclax will be administered orally
  Other Names: VENCLEXTA®; ME-522

SUMMARY:
This is a Phase 1, open-label, dose escalation study to determine the safety and preliminary efficacy of voruciclib monotherapy in subjects with relapsed/refractory B cell malignancies or AML after failure of standard therapies or voruciclib in combination with venetoclax in subjects with relapsed or refractory AML

DETAILED DESCRIPTION:
This is a Phase 1, open-label, 3 + 3 dose escalation and expansion study to determine the safety and preliminary efficacy of voruciclib monotherapy in subjects with relapsed/refractory B cell malignancies or AML after failure of prior standard therapies or voruciclib in combination with venetoclax in subjects with relapsed or refractory AML. Escalation to the next higher dose level will depend on demonstrated safety and tolerability at each dose level.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Histologically-confirmed diagnosis of Follicular lymphoma (FL), mantle cell lymphoma (MCL), marginal zone lymphoma (MZL), small lymphocytic lymphoma (SLL), chronic lymphocytic leukemia(CLL), diffuse large B-cell lymphoma (DLBCL), or AML

  a. Subjects must have disease that has relapsed or is refractory to 2 or more prior regimens and in need of treatment due to progressive disease
* Presence of measurable disease defined per the 2008 International workshop on CLL guidelines, or by 2014 Lugano criteria for non-Hodgkin lymphoma (does not apply for AML subjects)
* Adequate hematologic parameters unless clearly due to the disease under study
* Adequate renal and hepatic function, per laboratory reference range at screening

Exclusion Criteria:

* History of pneumonitis of any cause
* For CLL subjects: only known histological transformation to an aggressive lymphoma
* For AML subjects:

  1. Acute promyelocytic leukemia
  2. Peripheral blast count > 25 × 10 9/L
* Known central nervous system involvement
* Significant cardiovascular disease
* Significant screening ECG abnormalities
* Subjects who require warfarin, anti-cancer therapeutics or investigational agents
* Evidence of an ongoing systemic bacterial, fungal, or viral infection (including upper respiratory tract infections) at the time of start of voruciclib therapy
* Prior solid organ transplantation
* Receipt of an allogeneic transplant within 6 months or an autologous transplant within the preceding 3 months; evidence of ongoing graft-versus-host disease (GVHD)
* Prior therapy with a cyclin-dependent kinase (CDK9) inhibitor
* Symptomatic/uncontrolled HIV infection/AIDS, or currently taking contraindicated medications for HIV control
* Ongoing immunosuppressive treatment including calcineurin inhibitors at the time of the start of study treatment, including systemic or enteric corticosteroids except as follows:

  1. Prior to the start of study treatment, subjects may be using systemic corticosteroids (≤20 mg/day of prednisone or equivalent), topical, or inhaled corticosteroids
  2. During study therapy, subjects may use systemic, topical, or enteric corticosteroids, if needed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-05-31 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Determine the safety and tolerability of voruciclib | 2 years
  Safety will be measured by the incidence of all AEs and SAEs, timing, grade [CTCAE v4.03] severity, seriousness, relatedness.
  Tolerability will be measured by the incidence of DLTs (dose limiting toxicities)
Determine the safety and tolerability of voruciclib in combination with venetoclax in subjects with AML. | 2 years
  Safety will be measured by the incidence of all AEs and SAEs, timing, grade [CTCAE v4.03] severity, seriousness, relatedness.
  Tolerability will be measured by the incidence of DLTs (dose limiting toxicities)

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | 2 years
  defined as the sum of complete response (CR), complete remission with incomplete marrow recovery (CRi) and partial response (PR) for B-cell malignancies, or for AML the sum of CR/CRi rate by the 2017 European LeukemiaNet (ELN) criteria
Duration of Response (DOR) | 2 years
  defined as the time from the initial determination of response to the time of disease progression or death on study, which ever occurs first
Progression Free Survival (PFS) | 2 years
  defined as the time from the first dose of study drug administration (Cycle 1 Day 1) to disease recurrence or progression as defined by IWG criteria, or death on study
Evaluate the PK of voruciclib | 2 years
  Determined by the Area Under the Concentration time curve (AUC)
Evaluate the PK of voruciclib Cmax in combination with venetoclax Determined by the Area Under the Concentration time curve (AUC) | 2 years
  Determined by the Area Under the Concentration time curve (AUC)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - City of Hope, Duarte, California
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - New York University, New York, New York
  - Duke University, Durham, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - MD Anderson, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
  - Swedish Cancer Institute, Seattle, Washington
  - Froedtert Hospital & the Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Alvarado-Valero Y, Cook RJ, Dinner SN, Keng M, Begna KH, Javidi-Sharifi N, Abedin S, Al Malki MM, Bhatt VR, Rajagopalan P, Tang M, Wiley SE, Ghalie RG, Davids MS. The oral CDK9 inhibitor voruciclib combined with venetoclax for patients with relapsed/refractory acute myeloid leukemia. Blood Neoplasia. 2025 Apr 25;2(3):100108. doi: 10.1016/j.bneo.2025.100108. eCollection 2025 Aug. PMID 40809193
- [Derived] Davids MS, Brander DM, Alvarado-Valero Y, Diefenbach CS, Egan DN, Dinner SN, Javidi-Sharifi N, Al Malki MM, Begna KH, Bhatt VR, Abedin S, Cook RJ, Collins MC, Roleder C, Dominguez EC, Rajagopalan P, Wiley SE, Ghalie RG, Danilov AV. A phase 1 study of the CDK9 inhibitor voruciclib in relapsed/refractory acute myeloid leukemia and B-cell malignancies. Blood Adv. 2025 Feb 25;9(4):820-832. doi: 10.1182/bloodadvances.2024014633. PMID 39705540